CLINICAL TRIAL: NCT00247312
Title: Pd-103 Dose De-Escalation for Early Stage Prostate Cancer: A Prospective Randomized Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Schiffler Cancer Center (Other)
Responsible Party: Principal Investigator, Gregory Merrick, M.D., Medical Director, Schiffler Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 05-8-3
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Prostatic Neoplasm
Keywords: Prostate cancer; brachytherapy; palladium 103; I-125
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Palladium-103

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 125Gy prescription dose Pd-103 (Active Comparator): 125Gy prescription dose Pd-103
  Interventions: Radiation: Pd-103
- 110 Gy prescription dose Pd-103 (Active Comparator): 110 Gy prescription dose Pd-103
  Interventions: Radiation: Pd-103

INTERVENTIONS:
Radiation: Pd-103

SUMMARY:
The purpose of this study is to determine the most appropriate radiation implant dose for palladium-103 monotherapy. Radiation dose is related to potential cure. From previously published studies, it appears that the prescribed radiation dose can be reduced by 14-20% without any difference in potential cure (in this study, the dose is being decreased 10%). Although most patients tolerate brachytherapy well, complications to appear to be related to radiation exposure to normal structures (i.e. urethra, rectum and proximal penis). By reducing the prescribed dose, it is conceivable that fewer patients will experience side effects and complications.

DETAILED DESCRIPTION:
In calendar year 2003, approximately 220, 000 men will be diagnosed with prostate cancer and approximately 30,000 will die. The vast majority of men will be diagnosed with clinically organ-confined disease with potentially curative treatments including radical prostatectomy, external beam radiation therapy and brachytherapy. Within the uro-oncology community, the selection of one modality over another remains controversial.

Over the past decade, transperineal ultrasound-guided permanent prostate brachytherapy using either Pd-130 or I-125 has been increasingly utilized as definitive management for early stage carcinoma of the prostate gland. This resurgence of interest in prostate brachytherapy was the result of several technologic advances including the evolution of transrectal ultrasonography, the development of a closed transperineal approach and the availability of sophisticated treatment planning computers. These imaging and planning advances significantly improved the accuracy of seed placement. In addition, the advent of CT-based postoperative dosimetry in the early 1990's provided a unique opportunity to evaluate quality and proactively predict outcome and complications.

Prostate brachytherapy represents the ultimate 3-dimensional conformal therapy and permits dose escalation far exceeding other modalities. Following permanent prostate brachytherapy with or without supplemental external beam radiation therapy, favorable long term biochemical outcomes have been reported for patients with low, intermediate and high risk features with a morbidity profile that compares favorably with competing local modalities (1,2)2).

Although there is no definitive evidence suggesting that either Pd-103 or I-125 is more efficacious than the other in terms of cure or side effects/complications, preliminary results of a prospective randomized trial suggests that Pd-103 may be more "dose forgiving" than I-125 (3). Long-term results demonstrate cancer eradication is highly correlated with delivered radiation dose. To date, postoperative dosimetry has primarily been described in terms of V 100/150/200 (volume of the gland receiving 100%, 150% and 200% of the prescription dose) and the D90 (the dose delivered to 90% of the prostate gland). Following I-125 monotherapy, A D90 greater than or equal to 140 Gy (day 30 dosimetry) is required for optimal long-term biochemical control (4,5)4)5). A dose of 140 Gy represents 96% of the standard I-125 prescription dose (145 Gy). In contrast, following Pd-103 monotherapy, A D90 greater than or equal to 100 Gy (day 30 dosimetry) and a D90 greater than or equal to 108 Gy (median day 22 dosimetry) have been reported to predict optimal biochemical outcomes (6,7)6)7). These Pd-103 doses represent 80% and 86% of the standard monotherapy prescription dose (125 Gy). In addition, a prospective randomized trial demonstrated that coverage of 90% or more of the prostate by 124 Gy of Pd-103 yields 98% change of being cancer-free three years following treatment (3).

Because of some seed placement uncertainty, however, the pre-plans are designed to deliver a higher radiation dose than necessary to most of the prostate gland (8). Additionally, there is a variable amount of edema that occurs from the implant procedure, moving seeds farther away from each other, again requiring a higher planned dose than actually needed.

Delivered radiation dose is paramount to securing long-term freedom from biochemical progression. Previously Merrick and colleagues reported that postoperative dosimetric quality for Pd-103 and I-125 in terms of V 100/150/200 and D90 were independent of prostate size, isotope selection, radiation implant dose prescription, the use of supplemental external beam radiation therapy, neoadjuvant androgen deprivation therapy and patient age (8-12)8)9)10)11)12). These results demonstrate the dosimetric reproducibility of Pd-103 across all implant scenarios. A review of the last 200 consecutive Pd-103 implants at the Schiffler Cancer Center illustrates similar dosimetric outcomes for patients implanted with 125 Gy versus 115 Gy.

Although the morbidity profile of permanent prostate brachytherapy compares favorably with competing local modalities, side effects and complications do occur. Delivered radiation dose to the urethra, rectum and proximal penis strongly correlate with brachytherapy-related morbidity (2, 13-18)13)14)15)16)17)18).

In summary, the available literature suggests that the Pd-103 doses necessary for cure care substantially less than currently prescribed, postoperative dosimetry has consistently demonstrated high intraprostatic doses and brachytherapy-related morbidity is related to radiation doses to normal surrounding structures. As such, we proposed to conduct a prospective randomized trial evaluating the effect of a 12% reduction in prescription dose (125 Gy vs. 110 Gy) on the ultimate cure and complication rates for low risk prostate cancer (PSA greater than or equal to 10 ng/mL, Gleason score greater than or equal to 6 and clinical stage T1b-T2b). To assure that the dose is adequate, intraoperative and postoperative dosimetry will be performed. Intraoperative dose evaluation will allow additional seeds to be implanted if needed to achieve minimum required dose.

ELIGIBILITY:
Inclusion Criteria:

* Low risk patients: Gleason score less than or equal to 6, PSA less than or equal to 10 ng/mL and clinical stage T1b-T2b (2002 AJCC.
* An enzymatic prostatic acid phosphatase must be obtained prior to implantation.
* No pelvic external beam radiation therapy for either prostate cancer or other malignancies.
* Androgen deprivation therapy less than 4 month duration for size reduction is allowable.
* No surgical staging for prostate cancer.
* A minimum of 5 year life expectancy.
* No other invasive cancer diagnosis other than non-melanoma skin cancer within the last 5 years.

Exclusion Criteria:

* Exclusion criteria will be limited to patients who do not meet the above eligibility criteria.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2005-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
PSA determinations will be obtained 3 months following implantation and then every 6 months. | every 6 months after inital PSA done at 3 months.
  PSA determinations will be obtained 3 months following implantation and then every 6 months.
Androgen deprivation therapy will not be initiated unless the PSA exceeds 10 ng/mL or distant metastases are detected. | depends on outcome
  Androgen deprivation therapy will not be initiated unless the PSA exceeds 10 ng/mL or distant metastases are detected.

SECONDARY OUTCOMES:
Following brachytherapy, I-PSS will be obtained on months 1, 3, 6, 12, 18, 24, 36, 48, 60. | months 1, 3, 6, 12, 18, 24, 36, 48, 60.
  Following brachytherapy, I-PSS will be obtained on months 1, 3, 6, 12, 18, 24, 36, 48, 60.
Following brachytherapy, R-FAS will be obtained on months 12, 36 and 60. | months 12, 36 and 60.
  Following brachytherapy, R-FAS will be obtained on months 12, 36 and 60.
Following brachytherapy, IIEF will be obtained on months 12, 36 and 60. | months 12, 36 and 60.
  Following brachytherapy, IIEF will be obtained on months 12, 36 and 60.
Post implant quality of life evaluations will be forwarded to Dr. G. Merrick as appropriate. | as needed
  Post implant quality of life evaluations will be forwarded to Dr. G. Merrick as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory S. Merrick, MD, Principal Investigator — Schiffler Cancer Center, Wheeling, WV; Kent E. Wallner, MD, Study Chair — Department of Veterans Affairs, Seattle, WA
Locations (2):
- United States (2):
  - Radiation Oncology 174 Department of Veterans Affairs, Seattle, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia

REFERENCES:
- [Background] Merrick GS, Wallner KE, Butler WM. Permanent interstitial brachytherapy for the management of carcinoma of the prostate gland. J Urol. 2003 May;169(5):1643-52. doi: 10.1097/01.ju.0000035544.25483.61. PMID 12686802
- [Background] Merrick GS, Wallner KE, Butler WM. Minimizing prostate brachytherapy-related morbidity. Urology. 2003 Nov;62(5):786-92. doi: 10.1016/s0090-4295(03)00558-2. No abstract available. PMID 14624895
- [Background] Wallner K, Merrick G, True L, Sutlief S, Cavanagh W, Butler W. 125I versus 103Pd for low-risk prostate cancer: preliminary PSA outcomes from a prospective randomized multicenter trial. Int J Radiat Oncol Biol Phys. 2003 Dec 1;57(5):1297-303. doi: 10.1016/s0360-3016(03)01448-2. PMID 14630265
- [Background] Stock RG, Stone NN, Tabert A, Iannuzzi C, DeWyngaert JK. A dose-response study for I-125 prostate implants. Int J Radiat Oncol Biol Phys. 1998 Apr 1;41(1):101-8. doi: 10.1016/s0360-3016(98)00006-6. PMID 9588923
- [Background] Stock RG, Stone NN, Dahlal M, Lo YC. What is the optimal dose for 125I prostate implants? A dose-response analysis of biochemical control, posttreatment prostate biopsies, and long-term urinary symptoms. Brachytherapy. 2002;1(2):83-9. doi: 10.1016/s1538-4721(02)00017-x. PMID 15062175
- [Background] Kollmeier MA, Stock RG, Stone N. Biochemical outcomes after prostate brachytherapy with 5-year minimal follow-up: importance of patient selection and implant quality. Int J Radiat Oncol Biol Phys. 2003 Nov 1;57(3):645-53. doi: 10.1016/s0360-3016(03)00627-8. PMID 14529768
- [Background] Potters L, Cao Y, Calugaru E, Torre T, Fearn P, Wang XH. A comprehensive review of CT-based dosimetry parameters and biochemical control in patients treated with permanent prostate brachytherapy. Int J Radiat Oncol Biol Phys. 2001 Jul 1;50(3):605-14. doi: 10.1016/s0360-3016(01)01473-0. PMID 11395226
- [Background] Merrick GS, Butler WM. Modified uniform seed loading for prostate brachytherapy: rationale, design, and evaluation. Tech Urol. 2000 Jun;6(2):78-84. PMID 10798804
- [Background] Merrick GS, Butler WM, Dorsey AT, Lief JH. Potential role of various dosimetric quality indicators in prostate brachytherapy. Int J Radiat Oncol Biol Phys. 1999 Jun 1;44(3):717-24. doi: 10.1016/s0360-3016(99)00067-x. PMID 10348304
- [Background] Merrick GS, Butler WM, Dorsey AT, Lief JH. Effect of prostate size and isotope selection on dosimetric quality following permanent seed implantation. Tech Urol. 2001 Sep;7(3):233-40. PMID 11575521
- [Background] Merrick GS, Butler WM, Dorsey AT, Lief JH, Totterd, Coram RJ. Influence of prophylactic dexamethasone on edema following prostate brachytherapy. Tech Urol. 2000 Jun;6(2):117-22. PMID 10798812
- [Background] Merrick GS, Butler WM, Wallner KE, Galbreath RW, Adamovich E. Permanent interstitial brachytherapy in younger patients with clinically organ-confined prostate cancer. Urology. 2004 Oct;64(4):754-9. doi: 10.1016/j.urology.2004.04.054. PMID 15491715
- [Background] Merrick GS, Butler WM, Wallner KE, Galbreath RW, Lief JH. Long-term urinary quality of life after permanent prostate brachytherapy. Int J Radiat Oncol Biol Phys. 2003 Jun 1;56(2):454-61. doi: 10.1016/s0360-3016(02)04600-x. PMID 12738320
- [Background] Merrick GS, Butler WM, Tollenaar BG, Galbreath RW, Lief JH. The dosimetry of prostate brachytherapy-induced urethral strictures. Int J Radiat Oncol Biol Phys. 2002 Feb 1;52(2):461-8. doi: 10.1016/s0360-3016(01)01811-9. PMID 11872293
- [Background] Merrick GS, Butler WM, Wallner KE, Lief JH, Anderson RL, Smeiles BJ, Galbreath RW, Benson ML. The importance of radiation doses to the penile bulb vs. crura in the development of postbrachytherapy erectile dysfunction. Int J Radiat Oncol Biol Phys. 2002 Nov 15;54(4):1055-62. doi: 10.1016/s0360-3016(02)03031-6. PMID 12419431
- [Background] Herrmann RG, Bohnert HJ, Kowallik KV, Schmitt JM. Size, conformation and purity of chloroplast DNA of some higher plants. Biochim Biophys Acta. 1975 Jan 20;378(2):305-17. doi: 10.1016/0005-2787(75)90118-5. PMID 1092350
- [Background] Snyder KM, Stock RG, Hong SM, Lo YC, Stone NN. Defining the risk of developing grade 2 proctitis following 125I prostate brachytherapy using a rectal dose-volume histogram analysis. Int J Radiat Oncol Biol Phys. 2001 Jun 1;50(2):335-41. doi: 10.1016/s0360-3016(01)01442-0. PMID 11380219
- [Background] Merrick GS, Butler WM, Wallner KE, Hines AL, Allen Z. Late rectal function after prostate brachytherapy. Int J Radiat Oncol Biol Phys. 2003 Sep 1;57(1):42-8. doi: 10.1016/s0360-3016(03)00501-7. PMID 12909214
- [Background] Consensus statement: guidelines for PSA following radiation therapy. American Society for Therapeutic Radiology and Oncology Consensus Panel. Int J Radiat Oncol Biol Phys. 1997 Mar 15;37(5):1035-41. No abstract available. PMID 9169810